CLINICAL TRIAL: NCT00884936
Title: Identification of Gene Biomarkers in Aging Skin; a Blinded, Prospective, Single-center, Clinical Study
Brief Title: Identification of Gene Biomarkers in Aging Skin
Status: Completed | Type: Observational
Sponsor: Interleukin Genetics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ILI-08-112-USKAG
Record Dates: First submitted 2009-04-20; First posted 2009-04-21 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2009-10

CONDITIONS: Hyperpigmentation; Skin Aging
Keywords: Skin; Aging; Dermogenomics; Genetic; Biomarker; Dermatology
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 4 mm punch biopsy taken from exposed and unexposed skin.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Group 1: Young age: 20 to 30 years old
- Group 2: Middle Age: 38 to 48 years old (pre-menopausal only)
- Group 3: Elderly Age: 60 to 75 years old (Post-menopausal only)

SUMMARY:
This study is a blinded, prospective, single-center, clinical study conducted in Japanese female subjects between the ages of 20-75 years. This design uses skin biopsy samples from environmentally exposed areas and unexposed (control) areas within the same subjects to assess the gene expression profile from three different age groups.

DETAILED DESCRIPTION:
The primary objective of the skin aging study is to investigate changes in gene expression patterns that occur during the aging process.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are willing to read and sign an informed consent form prior to participating in the study.
* Individuals who have a temperature of less than or equal to 100 degrees F at the time of biopsy collection.
* Individuals who had not applied any sunless tanning product on the arms within the past year.
* Individuals with no prior history of alcoholism (or who consume fewer than 2 to 3 alcoholic beverages per day).
* Individuals who have not consumed any anti-aging nutritional supplements (multivitamins and multiminerals are acceptable) or aspirin, NSAIDS, or other pain medication in the last 48 hours before biopsy.

Exclusion Criteria:

* Male gender
* Individuals who did not fit the 'inclusion criteria' above.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asian female subjects between the ages of 20 to 75 years old who are non-smokers with no history of prior alcoholism.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2008-08; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to investigate changes in gene expression patterns that occur during the aging process. A significant fold change in differential gene expression will be >1.5 and an adjusted p-value of <0.05. | 1 year

SECONDARY OUTCOMES:
Secondary outcome measures are the evaluation of genetic expression changes in sun-protected and sun-exposed skin and an investigation of their biological pathways. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prakash Prabhakar, PhD, Study Director — Interleukin Genetics; Karen Shaver, MS, Study Director — Interleukin Genetics
Locations (1):
- Thomas J. Stephens & Associates, Japan Research Center, Tokyo, Japan